CLINICAL TRIAL: NCT00810953
Title: A Phase I/II Clinical Study Using Pentamidine in Patients With Locally Advanced or Metastatic Pancreatic Cancer Undergoing Standard Therapy
Brief Title: A Safety Study Using Pentamidine in Patients With Pancreatic Cancer Undergoing Standard Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncozyme Pharma Inc. (Industry)
Responsible Party: Dr. Terry Chow/President, Oncozyme Pharma Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-103-P
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pentamidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Use of pentamidine in locally advanced or metastatic pancreatic cancer
  Interventions: Drug: Pentamidine

INTERVENTIONS:
Drug: Pentamidine — two dose of 6 mg/kg with or without standard chemotherapy.

SUMMARY:
The purpose of this study is to investigate the safety and possible efficacy of the use of pentamidine in the treatment of pancreatic cancer metastasis in subjects receiving standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of advanced pancreatic adenocarcinoma that is unresectable or metastatic. At least one uni-dimensionally measurable lesion (on spiral CT scan)
* 18 years of age or older
* ECOG performance status 0, 1 or 2
* Serum aspartate transaminase (AST) serum alanine transaminase (ALT) £ 2.5 x upper limit of normal (ULN), or AST and ALT £ 5 x ULN if liver function abnormalities are due to underlying malignancy
* Total serum bilirubin £ 2 x ULN
* lipase within normal limits (1.5x ULN)
* Absolute neutrophil count (ANC) ≥ 1500/uL (1.5 x 109/L)
* Platelets ≥ 100,000/uL
* Hemoglobin ≥ 9.0 g/dL
* Serum creatinine £ 1.5 x ULN or calculated creatinine clearance ≥ 50 ml/min
* CA19-9 level ≥ 37 U/ml
* Normal ECG
* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrolment
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other trial procedures
* Life expectancy, in the opinion of the investigator, > 3 months

Exclusion Criteria:

* BP < 100 (systolic)
* History of uncontrolled renal disease, pancreatitis, or diabetes mellitus
* Peripheral sensory neuropathy (> Grade 1, as per NCI CTCAE version 3.0)
* Concomitant therapy with other investigational agents or participation in another clinical trial within the previous 3 months.
* Any of the following conditions: Ongoing cardiac dysrhythmias of NCI CTCAE grade ≥ 2; atrial fibrillation of any grade; QTc interval >450 msec for males or >470 msec for females or uncontrolled intercurrent illness, e.g., unstable angina; severe coronary disease, ventricular arrhythmias, bradycardia <50 bpm
* Active uncontrolled bacterial infection
* Concurrent use of drugs that could prolong QT interval
* Concurrent use of nephrotoxic drugs, including aminoglycosides, ampho B, foscarnet, cidofovir
* Concurrent use of drugs that may be associated with pancreatitis
* Concurrent active cancer originating from a primary site other than pancreas or history of cancer < 3 years except for skin superficial bladder, uterus etc
* History of allergy or hypersensitivity to pentamidine
* Pregnancy or breastfeeding. All female patients with reproductive potential must have a negative pregnancy test (serum or urine) prior to first dose of study medication.
* Severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgement of the investigator, excess risk associated with trial participation of study drug administration, or which in the judgement of the investigator, would make the subject inappropriate for entry into this trial.
* On oral anticoagulants (LMWH is acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Any severe events, tumor marker CA19-9, and tumor size (CT scan) | 6 months

SECONDARY OUTCOMES:
TDP | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Petr Kavan, MD, Ph.D., Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada